CLINICAL TRIAL: NCT00284921
Title: A Twelve-month, Randomized, Multicenter, Open-label, Exploratory Study to Investigate the Clinical Outcomes of an Immunosuppressive Regimen of Basiliximab, Cyclosporine Microemulsion (CsA-ME) and Enteric-coated Mycophenolate Sodium (EC-MPS) Free of Steroids Compared With a Regimen of EC-MPS With Standard Steroids in de Novo Kidney Recipients Who Are Hepatitis C Positive
Brief Title: MYPROMS-ES02: Safety and Efficacy of Basiliximab, Cyclosporine Microemulsion and Enteric-coated Mycophenolate Sodium (EC-MPS) Versus EC-MPS and Steroid Therapy in Kidney Transplant Recipients Who Are Hepatitis C Positive
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CERL080AES02
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: De Novo Kidney Transplant
Keywords: kidney transplant, hepatitis C, enteric-coated mycophenolate sodium
MeSH Terms: conditions — Hepatitis C

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS)

SUMMARY:
To prospectively evaluate in de novo kidney transplant recipients, hepatitis C positive, the clinical outcomes of an immunosuppressive regimen of EC-MPS free of steroids in comparison with a regimen of EC-MPS with standard steroids, as measured by the hepatic function tests (ALT/AST) after 12 months treatment.

ELIGIBILITY:
Inclusion criteria

1. Patients hepatitis C positive (serology test within the last 12 months and determined by third-generation assay).
2. Recipients of heart-beating cadaveric, living unrelated or living related non-HLA identical donor kidney transplant, treated with basiliximab and CsA-ME as primary immunosuppression.

Exclusion criteria

1. Multi-organ recipients (e.g. double kidney, kidney and pancreas or kidney and liver) or previous transplant with any other organ.
2. Kidneys from non-heart beating donors.
3. ABO incompatibility against the donor.
4. Patients with panel reactive antibodies of >50% at most recent assessment prior to transplantation and /or prior graft lost due to immunological reasons in the first six months post-transplantation or patients who are considered to be at increased risk of acute rejection by the principal investigator Additional protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-04; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Hepatic function tests (ALT/AST) after 12 months treatment.

SECONDARY OUTCOMES:
Acumulative incidence of biopsy proven acute rejection after 3 and 12 months.
Graft loss, biopsy-proven acute rejection after 3 and 12 months treatment.
Glomerular filtration rate and by proteinuria after 12 months treatment.
Graft survival after 12 months.
Incidence of AEs and SAEs after 3 and 12 months.
Blood pressure, lipids and glucose profiles after 3 and 12 months.
Percentage of patients free of steroids at 12 months between the two investigational groups.
Viral load (HCV RNA) between both groups at 12 months.
Bone density at 12 months in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis